CLINICAL TRIAL: NCT01310699
Title: Full Inspection With Narrow Band Imaging (NBI) for Detection of Flat Lesions And Tumors During Colonoscopy- The FIND FLAT Colonoscopy Study
Brief Title: Study of Flat Polyp Detection Using New Narrow Band Imaging (NBI) Compared to White Light Colonoscopy - The FIND FLAT Colonoscopy Study
Acronym: NBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Collaborators: Kansas City Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Roy Soetikno, Co-Principal Investigator, VA Palo Alto Health Care System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: FIND FLAT PA19624
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-10

CONDITIONS: Colorectal Neoplasms; Colonic Polyps; Colorectal Cancer
Keywords: Colonoscopy; Diagnostic imaging; Colorectal Neoplasm; Tandem Colonoscopy; Flat Polyp; Nonpolypoid; Flat and Depressed Lesions; Primary Prevention; Endoscopy
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Definition NBI Colonoscopy (Experimental): Use of high definition narrow band imaging colonoscopy during examination for polyp detection. The same intervention is used on both arms: the Olympus Colonoscope CFHQ190AL, a technically improved colonoscope with close focus high definition narrow band imaging.
  Interventions: Device: Olympus Colonoscope CFHQ190AL
- High Definition White Light Colonoscopy (Placebo Comparator): Use of high definition white light colonoscopy during examination for polyp detection. The same intervention is used on both arms: the Olympus Colonoscope CFHQ190AL, a technically improved colonoscope with close focus high definition narrow band imaging.
  Interventions: Device: Olympus Colonoscope CFHQ190AL

INTERVENTIONS:
Device: Olympus Colonoscope CFHQ190AL — Technically improved colonoscope with close focus high definition narrow band imaging.

SUMMARY:
We hypothesize that high definition narrow band imaging (NBI) colonoscopy compared to high definition white light colonoscopy will detect an increased number of nonpolypoid (flat and depressed) colorectal neoplasm.

DETAILED DESCRIPTION:
Interval colorectal cancers diagnosed within a three year period following a clearing colonoscopy have been reported at a rate of 1 cancer/1000 person years.The majority of these cancers are likely a consequence of a missed neoplastic lesion during routine colonoscopy. Recent tandem colonoscopy studies have shown no significant difference in adenoma miss or detection rates using narrow band imaging as compared to colonoscopy using white light. However, higher detection of flat neoplastic lesions using NBI was shown in a meta-analysis and should be furthered studied, especially considering that they are thought to be a strong contributor to a false negative colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients referred for routine colonoscopy are eligible

Exclusion Criteria:

* Known Inflammatory bowel disease
* Referred for endoscopic evaluation and removal of colorectal lesion
* Personal or family history of polyposis or non-polyposis syndrome
* Presentation for emergency endoscopy
* Inability to remove polyp due to coagulopathy or thrombocytopenia
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2013-01; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tonya Kaltenbach, MD MS, Principal Investigator — San Francisco Veterans Affairs Medical Center
Locations (3):
- United States (3):
  - Veterans Affairs Palo Alto, Palo Alto, California
  - Veterans Affairs San Francisco, San Francisco, California
  - Veterans Affairs Kansas City, Kansas City, Missouri

REFERENCES:
- [Background] Soetikno RM, Kaltenbach T, Rouse RV, Park W, Maheshwari A, Sato T, Matsui S, Friedland S. Prevalence of nonpolypoid (flat and depressed) colorectal neoplasms in asymptomatic and symptomatic adults. JAMA. 2008 Mar 5;299(9):1027-35. doi: 10.1001/jama.299.9.1027. PMID 18319413
- [Background] Kaltenbach T, Friedland S, Soetikno R. A randomised tandem colonoscopy trial of narrow band imaging versus white light examination to compare neoplasia miss rates. Gut. 2008 Oct;57(10):1406-12. doi: 10.1136/gut.2007.137984. Epub 2008 Jun 3. PMID 18523025
- [Background] Kaltenbach T, Soetikno R. Image-enhanced endoscopy is critical in the detection, diagnosis, and treatment of non-polypoid colorectal neoplasms. Gastrointest Endosc Clin N Am. 2010 Jul;20(3):471-85. doi: 10.1016/j.giec.2010.04.001. PMID 20656245
- [Background] Rex DK, Bond JH, Feld AD. Medical-legal risks of incident cancers after clearing colonoscopy. Am J Gastroenterol. 2001 Apr;96(4):952-7. doi: 10.1111/j.1572-0241.2001.03677.x. PMID 11316211
- [Background] Rex DK, Helbig CC. High yields of small and flat adenomas with high-definition colonoscopes using either white light or narrow band imaging. Gastroenterology. 2007 Jul;133(1):42-7. doi: 10.1053/j.gastro.2007.04.029. Epub 2007 Apr 20. PMID 17631129
- [Background] van den Broek FJ, Reitsma JB, Curvers WL, Fockens P, Dekker E. Systematic review of narrow-band imaging for the detection and differentiation of neoplastic and nonneoplastic lesions in the colon (with videos). Gastrointest Endosc. 2009 Jan;69(1):124-35. doi: 10.1016/j.gie.2008.09.040. No abstract available. PMID 19111693

RESULTS

PARTICIPANT FLOW:
Groups:
- High Definition NBI Colonoscopy: Use of high definition narrow band imaging colonoscopy during examination for polyp detection.
  Olympus Colonoscope CFHQ190AL: Technically improved colonoscope with close focus high definition narrow band imaging.
- High Definition White Light Colonoscopy: Use of high definition white light colonoscopy during examination for polyp detection.
  Olympus Colonoscope CFHQ190AL: Technically improved colonoscope with close focus high definition narrow band imaging.
Period: Overall Study
Arm/Group | High Definition NBI Colonoscopy | High Definition White Light Colonoscopy
Started | 132 | 149
Completed | 128 | 143
Not Completed | 4 | 6
Not completed — Patients did not complete tandem. | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Definition NBI Colonoscopy | High Definition White Light Colonoscopy | Total
Number analyzed (Participants) | 128 | 143 | 271
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (9.4) | 62.3 (8.6) | 63 (9.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 11
  Male | 125 | 135 | 260

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Nonpolypoid (Flat and Depressed) Colorectal Neoplasm
Description: Compare the nonpolypoid colorectal neoplasm detection characteristics of the new high definition narrow band imaging colonoscopy to conventional high definition white light mode colonoscopy.
Time Frame: One week (time of procedure plus time for pathology of polyp to be analyzed by histology)
Measure: Count of Participants; unit: Participants
Arm/Group | High Definition NBI Colonoscopy | High Definition White Light Colonoscopy
Number analyzed (Participants) | 128 | 143
Participants | 33 | 43

2. Secondary Outcome: Percentage of Missed Lesions on Index Colonoscopy.
Description: Compare the number of missed lesions on the index examination using the new high definition narrow band imaging colonoscopy to the conventional high definition white light mode colonoscopy, based on the tandem colonoscopy findings.
Time Frame: One week (time of procedure plus time for pathology of polyp to be analyzed by histology)
Measure: Number; unit: percentage of adenomas
Arm/Group | High Definition NBI Colonoscopy | High Definition White Light Colonoscopy
Number analyzed (Participants) | 128 | 143
percentage of adenomas | 32.0 | 31.4
Statistical Analysis 1: Comparison: High Definition NBI Colonoscopy vs High Definition White Light Colonoscopy; Test type: Superiority; p = 0.21, Chi-squared

3. Secondary Outcome: Percentage of Nonpolypoid (Flat) Missed Lesions
Description: Compare the number of missed non-polypoid lesions on the index examination using the new high definition narrow band imaging colonoscopy to the conventional high definition white light mode colonoscopy.
Time Frame: One week (time of procedure plus time for pathology of polyp to be analyzed by histology)
Population: Adenoma by shape (i.e. Flat)
Measure: Number; unit: percentage of adenomas
Arm/Group | High Definition NBI Colonoscopy | High Definition White Light Colonoscopy
Number analyzed (Participants) | 128 | 143
percentage of adenomas | 7.2 | 11.8
Statistical Analysis 1: Comparison: High Definition NBI Colonoscopy vs High Definition White Light Colonoscopy; Test type: Superiority; p = 0.18, Chi-squared

ADVERSE EVENTS:
Arm/Group | High Definition NBI Colonoscopy | High Definition White Light Colonoscopy
Serious Adverse Events (participants affected / at risk) | 0/128 | 0/143
Other Adverse Events (participants affected / at risk) | 0/128 | 0/143

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No